CLINICAL TRIAL: NCT03431701
Title: Chlorhexidine Vaginal Cleansing Versus Iodine Prior to C-section and the Rate of Postoperative Infection: Randomized Clinical Trial
Brief Title: Chlorhexidine Vaginal Cleansing Versus Iodine Prior to C-section and the Rate of Postoperative Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Manal Hubeish, OBGYN attending physician, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 01022018
Record Dates: First submitted 2018-02-05; First posted 2018-02-13 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Vaginal Scrubbing
MeSH Terms: interventions — Chlorhexidine; Iodine; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group chlorhexidine (Experimental): Patients will receive chlorhexidine abdominal and vaginal scrubbing
  Interventions: Other: Chlorhexidine; Other: Antibiotics
- Group iodine (Active Comparator): Patients will receive iodine abdominal and vaginal scrubbing
  Interventions: Other: Iodine; Other: Antibiotics

INTERVENTIONS:
Other: Chlorhexidine — Vaginal cleansing will be performed in conjunction with the abdominal preparation with foam sponge that contains chlorhexidine. A sponge soaked with chlorhexidine will be inserted into the vagina and rotated 360 degrees in the vaginal cavity for about 30 seconds
  Arms: Group chlorhexidine
Other: Iodine — Vaginal cleansing will be performed in conjunction with the abdominal preparation with foam sponge that contains iodine. A sponge soaked with iodine will be inserted into the vagina and rotated 360 degrees in the vaginal cavity for about 30 seconds
  Arms: Group iodine
Other: Antibiotics — All participants will receive a single body mass index (BMI) based antibiotic dose of cefazolin or clindamycin within 30 minutes prior to the incision.

SUMMARY:
Background: Women undergoing cesarean delivery have 5 to 20 fold greater risk for infection and infectious morbidity compared with those undergoing vaginal birth. Endometritis, febrile morbidity, and wound infection are the most frequent complications of post cesarean infections. Endometritis accounts for 6-27% followed by clinically significant fever, which was reported about 5-24%,while the incidence of wound infection is about 2-9%.Previous studies evaluated whether vaginal cleansing can reduce the incidence of postoperative infectious morbidity. In most of the studies, povidone iodine was used as intervention.

Objectives: The aim of this study is to test the hypothesis that preoperative vaginal cleansing with chlorhexidine would be superior to iodine for the prevention of maternal infectious morbidities including endometritis, fever and wound complications.

Methods: This prospective randomized single blinded controlled trial will be conducted at Makassed General Hospital between February 2018 and January 2019. Total of 300 patients, 150 in each group, will be enrolled. Group 1 patients will receive chlorhexidine vaginal cleansing while group 2 patients will receive iodine prior to C-section. Adverse post infectious morbidities such as endometritis, febrile illness and wound infections will be observed within 30 days of C-section.

DETAILED DESCRIPTION:
This prospective randomized single blinded controlled trial will be conducted at Makassed General Hospital between February 2018 and January 2019. All pregnant women who will undergo cesarean delivery and willing to sign the informed consent will be included. Total of 300 patients, 150 in each group, will be enrolled. Group 1 patients will receive chlorhexidine vaginal cleansing while group 2 patients will receive iodine prior to C-section. Adverse post infectious morbidities such as endometritis, febrile illness and wound infections will be observed d within 30 days of C-section.

Vaginal cleansing will be performed in conjunction with the abdominal preparation with foam sponge that contains either chlorhexidine or iodine, sponge will be inserted into the vagina and rotated 360 degrees in the vaginal cavity for about 30 sec. All participants will receive a single body mass index (BMI) based antibiotic dose of cefazolin within 30 minutes prior to the incision.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women who will undergo cesarean delivery
* and willing to sign the informed consent.

Exclusion Criteria:

* Known allergy to the antiseptics used
* Infection diagnosis on admission
* Age ≤ 17 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Infectious morbidities | Within 30 days
  post cesarean infectious morbidities: endometritis, febrile morbidity and wound infection

SECONDARY OUTCOMES:
Length of hospital stay | Within 30 days
  Length of hospital stay after delivery
Readmission to the hospital | Within 30 days
  Percentage of patients readmitted to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hubesih, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon